CLINICAL TRIAL: NCT01673438
Title: An Open-Label Phase 1b Study to Investigate the Safety and Maximum Tolerated Dose of Aldoxorubicin (INNO-206) Plus Doxorubicin HCL Administered as Infusions Every 3 Weeks in Subjects With Advanced Solid Tumors
Brief Title: Phase 1b Study to Investigate the Safety and Maximum Tolerated Dose of Aldoxorubicin (INNO-206) Plus Doxorubicin HCL in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALDOXORUBICIN-P1-MTD-02
Record Dates: First submitted 2012-08-21; First posted 2012-08-28 (Estimated); Last update posted 2022-02-10 (Actual); Status verified 2014-04

CONDITIONS: Advanced Solid Tumor
Keywords: solid tumor; aldoxorubicin; phase 1; INNO-206; doxorubicin
MeSH Terms: interventions — DOXO-EMCH

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aldoxorubicin plus doxorubicin (Experimental): Aldoxorubicin dosages of 175, 240, and 320 (doxorubicin equivalents of 130, 180, and 240 mg/m2) will be administered as a 30 minutes IVI on Day 1 of each cycle. In addition 35 mg/m2 of doxorubicin HCl will be administered as an IVI over > 3 minutes no later than 3 hours, but no more than 6 hours before the start of aldoxorubicin infusion.
  Interventions: Drug: aldoxorubicin

INTERVENTIONS:
Drug: aldoxorubicin
  Other Names: INNO-206

SUMMARY:
This is a phase 1b open-label study to investigate the safety and maximum tolerated dose of aldoxorubicin plus doxorubicin HCl adminstered as infusion every 3 weeks for up to 8 cycles in subjects with advance solid tumors.

DETAILED DESCRIPTION:
An Open-Label Phase 1b Study to Investigate the Safety and Maximum Tolerated Dose of Aldoxorubicin (INNO-206) Plus Doxorubicin HCl Administered as Infusions Every 3 Weeks in Subjects with Advanced Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, male or female.
2. Histologically or cytologically confirmed malignant solid tumor that has relapsed or is refractory to standard therapy or no standard chemotherapy exists.
3. Capable of providing informed consent and complying with trial procedures.
4. Baseline absolute left ventricular ejection fraction (LVEF) measured scintigraphically (MUGA, myocardial scintigram) or by ultrasound (echocardiogram) ≥ Institutional Lower Limit of Normal.
5. Eastern Cooperative Oncology Group performance status (ECOG PS) 0-2.
6. Life expectancy > 12 weeks.
7. Measurable or evaluable disease according to RECIST 1.1 criteria.15
8. Women must not be able to become pregnant (e.g., post-menopausal for at least 1 year, surgically sterile, or practicing adequate birth control methods) for the duration of the study. [Adequate contraception includes: oral contraception, implanted contraception, intrauterine device implanted for at least 3 months, or barrier method in conjunction with spermicide.]
9. Women of child bearing potential must have a negative serum or urine pregnancy test at the Screening Visit and be non-lactating.
10. Geographic accessibility to the site that ensures that the subject will be able to keep all study-related appointments.

Exclusion Criteria:

1. Palliative surgery, chemotherapy, immunotherapy and/or radiation treatment < 4 weeks prior to the Screening Visit.
2. Prior treatment with ≥ 150 mg/m2 doxorubicin HCl or Doxil® cumulative dose, or epirubicin ≥ 150 mg/m2.
3. Exposure to any investigational agent within 30 days of Randomization.
4. Evidence of active or uncontrolled central nervous system (CNS) metastasis (negative imaging study performed due to suspicion of CNS metastasis within 4 weeks of Screening Visit).
5. History of other malignancies except cured basal cell carcinoma, squamous cell carcinoma, superficial bladder cancer or carcinoma in situ of the cervix.
6. Laboratory values: Screening serum creatinine ≥ 2 times the upper limit of normal (ULN), alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 times the ULN if no liver metastases or 5 times the ULN if liver metastases, total bilirubin > 2 times the ULN, white blood cell (WBC) count < 3500/mm3, or absolute neutrophil count (ANC) < 1500/mm3, platelet concentration < 100,000/mm3, hematocrit level < 25% for females or < 27% for males, or coagulation tests (prothrombin time [PT]; partial thromboplastin time [PTT]), International Normalized Ration (INR) > 1.5 times the ULN, serum albumin < 2.0g/dL.
7. Clinically evident congestive heart failure (CHF) > class II of the New York Heart Association (NYHA) guidelines.
8. Baseline QTc > 470 msec and/or previous history of QT prolongation while taking other medications. Concomitant use of medications associated with a high incidence of QTc prolongation is not allowed.
9. Serious clinically significant cardiac arrhythmias, defined as the existence of an absolute arrhythmia or ventricular arrhythmias classified as Lown III, IV or V.
10. History or signs of active coronary artery disease with or without angina pectoris.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | up to 6 months
  The primary objective of this study is to determine the preliminary safety and maximum tolerated dose (MTD) of aldoxorubicin plus doxorubicin HCl in subjects with advanced solid tumors who have failed standard therapies.

SECONDARY OUTCOMES:
Tumor Response | up to 6 months
  The secondary objective of this study is to evaluate the tumor response to aldoxorubicin plus doxorubicin HCl in this population assessed by radiographic means using the RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Levitt, MD, Study Director — CytRx Coorporation
Locations (1):
- Sarcoma Oncology Center, Santa Monica, California, United States